CLINICAL TRIAL: NCT02188628
Title: Refinement and Clinical Evaluation of the H-Man: A Novel, Portable, Inexpensive Planar Robot for Arm Rehabilitation After Stroke
Brief Title: Refinement and Clinical Evaluation of the H-Man for Arm Rehabilitation After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Principal Investigator, Chua Sui Geok, Karen, Senior Consultant, Tan Tock Seng Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2014/00122
Record Dates: First submitted 2014-07-02; First posted 2014-07-11 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Stroke
Keywords: Motor recovery, robotics, stroke rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: H-Man training + conventional therapy vs equal amount of conventional therapy 1:1 allocation
Who Masked: Outcomes Assessor
Masking Description: Blinded therapist assessor to determine clinical outcomes at pre and post treatment and follow up.
Oversight: Data Monitoring Committee: No

ARMS (2):
- H-Man (Experimental): H-Man is a novel, portable, inexpensive end-effector upper limb robot.
  Interventions: Device: H-Man
- Additional Conventional Therapy (Active Comparator): Repetitive goals based arm therapy
  Interventions: Other: Additional Conventional Therapy

INTERVENTIONS:
Device: H-Man — H-man is a portable end-effector planar upper limb robot.
  Other Names: No other names.
  Arms: H-Man
Other: Additional Conventional Therapy — Repetitive goals based arm therapy
  Other Names: No other names
  Arms: Additional Conventional Therapy

SUMMARY:
Locally, stroke remains the 4th cause of death, causing 8.4% of deaths annually in Singapore, and a leading cause of neurological disability worldwide. Nearly 40% of the stroke survivors will require specialized rehabilitation. In recent years, robot-aided therapy has been proposed as a means of complementing traditional therapy to alleviate the burden on therapists and on the healthcare system. For shoulder/elbow rehabilitation, dozens of robots have been proposed in the literature but only half a dozen have been commercialized and typically none are seen in local clinics, due to exceedingly high costs. A novel, compact, inexpensive robotic interface, named 'H-Man', was recently designed and developed at NTU for experiments in motor control neuroscience. The H-man can generate computer-controlled force fields to assist or resist a subject's motion and is potentially an optimal trade-off between clinical efficacy and robotic complexity. A first prototype of the H-Man is available at NTU.The primary aim of this proposed project is to assess to what extent the investigators H-Man is suitable for rehabilitation purposes using a feasibility pilot clinical trial design involving stroke survivors. The investigators believe that H-Man can be used for neuro-rehabilitation of stroke patients with hemiparetic weakness, motor incoordination and motor ataxia of the upper limbs.In close cooperation between clinicians at the TTSH and NTU engineers, a portable version of the H-Man will be developed which will be tested in a 12 subject Pilot study, refined and then used in a 44 subject Randomized Controlled Trial (RCT) study. At the same time, the feasibility of H-Man integration for a pared down home use model will be assessed in 4 subjects.

The investigators primary hypothesis is that sub-acute/chronic patients will exhibit clinically significant decreases of impairment when training with the H-Man combined with standard arm therapy on robot-measured scales and standardized clinical scales, at the level of elbow/shoulder after 18 sessions of training on the H-Man.

DETAILED DESCRIPTION:
As above

ELIGIBILITY:
Inclusion Criteria:

* First ever clinical stroke (ischaemic or haemorrhagic) confirmed on brain imaging
* Duration post stroke: 3 months to 24 months
* Age 21 to 85 years
* Hemiplegic pattern of arm motor impairment with Shoulder abduction MRC motor power >/= 3/5 and elbow flexion MRC motor power >/= 3/5
* Affected upper limb Fugl Myer Motor Assessment (FMMA) scale 20-50
* And / or associated motor incoordination or motor ataxia

Exclusion Criteria:

* Non stroke related causes of arm motor impairment
* Medical conditions incompatible with research participation: uncontrolled medical illnesses (hypertension or diabetes, heart failure, asthma, depression, end stage renal failure, terminal malignancy), life expectancy <6 months, unhealed fractures or severe arm pain (visual analogue scale VAS > 5/10, pregnancy
* Inability to tolerate sitting for 90 minutes.
* Local factors which preclude robotic interfacing or may be worsened by intensive arm therapy: spasticity of Modified Ashworth Scale grades 3-4, skin wounds, shoulder pain VAS >5/10, active fractures or arthritis or fixed flexion contractures of shoulder, elbow, wrist or fingers incompatible with interface with the H-man robot.
* Severe sensory impairment of affected limb
* Severe visual impairment, hemispatial neglect or homonymous hemianopia
* Cognitive impairments or uncontrolled behaviour. (Folstein mini mental state exam MMSE <26/28)

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Fugl Meyer Assessment of Motor Recovery | 0, 3, 6, 12 and 24 weeks after start of intervention
  As above

SECONDARY OUTCOMES:
Change from Baseline in Action Research Arm Test | 0, 3, 6, 12 and 24 weeks after start of intervention
  As above

CONTACTS AND LOCATIONS:
Overall Officials: Chua SG Sui Geok, MBBS,FRCP, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Rehabilitation Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Budhota A, Chua KSG, Hussain A, Kager S, Cherpin A, Contu S, Vishwanath D, Kuah CWK, Ng CY, Yam LHL, Loh YJ, Rajeswaran DK, Xiang L, Burdet E, Campolo D. Robotic Assisted Upper Limb Training Post Stroke: A Randomized Control Trial Using Combinatory Approach Toward Reducing Workforce Demands. Front Neurol. 2021 Jun 2;12:622014. doi: 10.3389/fneur.2021.622014. eCollection 2021. PMID 34149587